CLINICAL TRIAL: NCT00839943
Title: Effect Of Obesity On Ozone-Induced Airway Inflammation
Acronym: OBOZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 05-CEMLB-128; IRB 05-1644
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: ozone; clean air
MeSH Terms: conditions — Obesity | interventions — Ozone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ozone (Active Comparator): obese vs non-obese women
  Interventions: Other: ozone, 0.4 ppm
- air (Active Comparator): obese vs non obese women
  Interventions: Other: ozone, 0.4 ppm

INTERVENTIONS:
Other: ozone, 0.4 ppm — 2 hour ozone exposure, 0.40 ppm

SUMMARY:
The purpose of this study is to compare the effect of ozone exposure on airway reactivity and inflammation in obese vs. non-obese adults.

DETAILED DESCRIPTION:
Obesity has been shown to be associated with initial onset of asthma in children and increased airway hyperresponsiveness in adults (1,2). An important aspect of these epidemiologic data is that the impact of obesity on asthma is much stronger in females than males. For example, the incidence of asthma after the age of 11 years is five- to sevenfold higher in female children who become obese versus those who remain lean, whereas no such relationship exists for males (3). Recent mouse models of obesity suggest that this condition enhances airway responses to ozone air pollution (4). These mice eat excessively due to a defect in the gene encoding leptin, a satiety hormone produced in adipocytes. Shore et al (4) showed that these leptin-deficient obese mice had greater airway hyperreactivity to i.v. methacholine following ozone exposure compared to lean, wild-type mice. Furthermore, administration of exogenous leptin (which is actually increased in the serum of obese individuals (4)) was shown to enhance ozone-induced cytokine and protein release into BAL fluid of lean, wild type mice (4). Reduced lung volumes and altered breathing patterns in the obese may also contribute to enhanced airway reactivity in these patients (5). Stretch of airway smooth muscle during tidal breathing and especially during deep breaths, i.e. sighs, acts as a potent bronchodilator that might ameliorate ozone-induced bronchoconstriction. The increased chest load associated with obesity may also diminish tidal breathing volumes and frequency of sighs during ozone exposure.

ELIGIBILITY:
Inclusion Criteria:

* Twenty (20) non-obese, non-overweight (body mass index, 18 kg/m2 > BMI < 25 kg/m2, waist circumference < 35 inches) subjects and 20 obese (30 kg/m2 > BMI < 38 kg/m2, waist circumference >= 35 inches) volunteer females between 18-35 yrs of age

Exclusion Criteria:

* Are female and pregnant or have any reason to believe you might be pregnant.
* Are not between 18 and 35 years old.
* Have a history of asthma or have current hay fever.
* Have ever smoked more than 10 cigarettes (one half pack) a month or smoked during the past 30 days.
* Have a history of acute or chronic cardiovascular disease, chronic respiratory disease, and acute respiratory illness within 4 weeks.
* Have contraindications for performing sustained light exercise.
* You've been in a recent or recurring exposure to a dusty environment at work
* If you are unwilling to refrain from strenuous physical activity for 24 hours before and after each exposure.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Methacholine reactivity (primary endpoint) | 2-4 hours post exposure

SECONDARY OUTCOMES:
Breathing and lung function variables | immediately post exposure, 24 post exposure
induced sputum markers | 4 hours post exposure

CONTACTS AND LOCATIONS:
Overall Officials: William Bennett, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Stephanie London, MD, PhD, Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- US EPA Human Studies Facility-UNC -CH campus, Chapel Hill, North Carolina, United States